CLINICAL TRIAL: NCT03762707
Title: Correlation Between Platelet Function Analyzer-100 Testing and Bleeding Events After Percutaneous Kidney Biopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: Prof. Carlo Manno (Unknown); Dott. Francesco Pesce (Unknown); Dott. Michele Rossini (Unknown); Dott. Vincenzo Di Leo (Unknown)
Responsible Party: Principal Investigator, Loreto GESUALDO, Full Professor of Nephrology, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Other Study IDs: LGPFA100
Record Dates: First submitted 2018-12-02; First posted 2018-12-04 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Blood Platelet Disorder; Hemorrhage; Kidney Diseases
Keywords: Platelet Function Analyser-100 (PFA-100); Kidney biopsy; Bleeding Complications
MeSH Terms: conditions — Blood Platelet Disorders; Hemorrhage; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Kidney biopsy represents the criterion standard to obtain information on diagnosis and prognosis of renal dysfunctions . Many patients with kidney disease have a predisposition to bleed, especially when they undergo an invasive procedure such as renal biopsy. The predominant factor is abnormal platelet function. Therefore, the aim of this study is to evaluate whether the platelet function analyzer (PFA-100), a very reliable test to investigate primary hemostasis, can be useful in predicting the risk of bleeding complications in patients undergoing renal biopsy.

DETAILED DESCRIPTION:
Kidney biopsy frequently is used to investigate the cause of suspected renal parenchymal disease. Although kidney biopsy may provide important diagnostic information and guide therapeutic decisions, the benefits must be weighed against the potential harms of biopsy. Bleeding is one of the most feared risks from a renal biopsy.

The technique has significantly evolved because of the introduction of real-time ultrasound guidance and use an automated spring-loaded biopsy device. As a consequence, the general safety and complication rate of the procedure has substantially improved. Post biopsy bleeding (hematoma and hematuria) is the primary complication of renal biopsies. However, most of the perirenal hematomas are minor and without clinical significance, and major complications are infrequent.

To minimize bleeding risk, we used the following prebiopsy parameters as a guide: prothrombin time (PT), activated partial thromboplastin time (aPTT), platelet count, age, sex, glomerular filtration rate and blood pressure. Antiaggregant and anticoagulant were stopped for 7 -10 days before biopsy. The Ivy bleeding time (BT) was performed.

Although an specific lancet is used to deliver a relatively standardized incision on the patient's forearm, the Ivy bleeding time technique is patient and operator-dependent. Skin thickness varies not only with age, but also with a number of other factors, such as nutritional status. For these reasons was developed the platelet function analyzer, PFA-100. This test assess primary haemostasis in vitro using citrated whole blood. The device simulates in vivo haemostatic plug formation under high shear flow by measuring the time required to occlude (closure time, CT) a collagen/epinephrine (Coll-EPI) or collagen/ADP (Coll-ADP)-coated aperture inserted in a plastic membrane. PFA-100 is more sensitive than BT to abnormalities of primary haemostasis.

The objective of this study is to demonstrate whether an abnormal PFA-100 can predict bleeding events after percutaneous kidney biopsy.

The present cohort includes 250 all adult patients who underwent percutaneous renal biopsy of native kidney in the Department of Emergency and Organ Transplantation, the University of Bari, Italy, from January 2017 to December 2018. Transplant kidney biopsies were excluded from this study. Three experienced nephrologists performed all the biopsies.

Participation included clinical data collection, serial blood and urine sampling before and after the procedure. Kidney ultrasound was performed in all patients before the procedure.

The following data were collected for all patients:

* Variables pre-biopsy:

  * baseline demographics (age, gender);
  * indication for renal biopsy [urinary abnormalities (i.e., proteinuria and haematuria), and/or recurrent macrohaematuria and/or nephrotic syndrome and/or nephritic syndrome and/or alteration of renal function and/or acute renal failure];
  * baseline systolic and diastolic blood pressure;
  * which kidney was biopsied;
  * baseline serum creatinine, azotaemia and glomerular filtration rate;
  * baseline haemoglobin and platelet count;
  * baseline coagulation parameters (prothrombin time, partial thromboplastin time, bleeding time);
  * baseline urinary protein excretion;
  * body mass index.
* Variables during-biopsy:

  * administration of DDAVP;
  * number of passes;
  * number of renal biopsy samples;
  * the position of the patient during kidney biopsy [prone position or supine anterolateral position (SALP)];
* Variables post-biopsy:

  * hemoglobin;
  * post-biopsy bleeding complications (gross hematuria, hematoma);
  * if was necessary transfusion of blood products or an invasive procedure (angiography and arterial embolization or surgery).

Evaluation of kidneys conditions were performed by ultrasound before the procedure in all patients. Longitudinal and transverse size, corticomedullary differentiation shape, location and related structures of the kidney were assessed using ultrasound and blood flow of the kidneys were assessed using a color-flow Doppler signal.

All biopsies were performed using real-time ultrasound-fixed guidance by a nephrologist with assistance from an expert in renal ultrasonography. A 16-gauge automated spring-loaded gun was used for the biopsy. A pathologist promptly examined the biopsy specimen under alight microscope to confirm that adequate renal tissue was available for further pathological evaluations. 1-deamino-8-D-arginine vasopressin (DDAVP) was administered to all patients who had not contraindication.

After the procedure, patients were invited to rest in bed on their backs for a 24-hour observation time. Meantime, clinical evaluation (gross haematuria, flank pain, hypotension) was performed to identify a bleeding complications. Ultrasound evaluation was performed for all patients after 24 hours from percutaneous renal biopsy to exclude a presence of complication, as hematoma and arteriovenous fistula Post biopsy bleeding complications were categorized as either minor or major. Minor bleeding complications included gross haematuria and/or subcapsular perinephric hematoma (<5cm diameter) that spontaneously resolved without need for further intervention. Major complications were defined as those that required an intervention for resolution, either the transfusion of blood products or an invasive procedure (angiography, surgery), and those that led to acute renal obstruction or failure, septicaemia, or death. The size of post biopsy hematoma (surface area) was defined as the product of the longest and the shortest diameters on the two-dimensional sonographic pictures.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing standard percutaneous renal biopsy performed in our Unit

Exclusion Criteria:

* contraindication to standard percutaneous renal biopsy

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The present cohort includes 250 all adult patients who underwent percutaneous renal biopsy of native kidney in the Department of Emergency and Organ Transplantation, the University of Bari, Italy, from January 2017 to December 2018. Transplant kidney biopsies were excluded from this study.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding After Kidney Biopsy | 24 hours
  Gross haematuria and/or subcapsular perinephric hematoma at ultrasound evaluation. Need for transfusion of blood products or an invasive procedure (angiography, surgery).

SECONDARY OUTCOMES:
Hemoglobin After Kidney Biopsy | 24 hours
  Anemization After Kidney Biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- AOUConsorziale Policlinico Di Bari, Bari, Italy